CLINICAL TRIAL: NCT03884530
Title: Ticagrelol Versus Aspirin in Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed zeinhom Gomaa, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2388
Record Dates: First submitted 2019-03-08; First posted 2019-03-21 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Acute Stroke; Ischemic Stroke
Keywords: ticagrelol; aspirin
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 2 groups. The first group formed of 85 patients will receive 180 mg ticagrelor (2 tablets of 90 mg) as a single loading oral dose and continue on 180 mg ticagrelor (1 tablet of 90 mg every 12 hours). The second group formed of 84 patients will receive 300 mg Aspirin (4 tablets of 75 mg) as a single loading oral dose, and will then be commenced on 300 mg Aspirin daily for 2 weeks then 75 mg daily after that. If the patients showed complications of the loading dose of ticagrelor (central or peripheral bleeding the dose will be minimized to 90 mg (1 tablet of 90 mg).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor ( Brilique) group (Active Comparator): the group will receive 180 mg ticagrelor (2 tablets of 90 mg) as a single loading oral dose, and continue on 180 mg ticagrelor (1 tablet of 90 mg every 12 hours) for 3 months
  Interventions: Drug: Ticagrelor (Brilique) 90
- Aspirin Group (Active Comparator): The group will receive 300 mg Aspirin (4 tablets of 75 mg) as a single loading oral dose, and will then be commenced on 300 mg Aspirin daily for 2 weeks then 75 mg daily after that for 3 months
  Interventions: Drug: Aspirin 75mg

INTERVENTIONS:
Drug: Ticagrelor (Brilique) 90 — Drug name Brilique 90 ml Drug form tablet
  Arms: Ticagrelor ( Brilique) group
Drug: Aspirin 75mg — Drug name Aspirin 75 ml Drug form tablet
  Arms: Aspirin Group

SUMMARY:
There is a debate whether ticagrelor is superior to aspirin in treating patients with ischemic stroke or not, most of the studies examine the effect of both drugs within 24 hours of acute stroke some find that there is no difference between ticagrelor and aspirin, others find that ticagrelor is superior to aspirin.

At this study the investigators aim at evaluating the role of loading ticagrelor received within 9 hours of acute ischemic stroke in improving neurological outcome of stroke. And evaluating the risk of hemorrhagic and non- hemorrhagic complications associated with the use of ticagrelor180 ml oral loading dose within 9 hours acute ischemic stroke

DETAILED DESCRIPTION:
ticagrelor is acyclo-pentyltriazolo-pyrimidine antiplatelet drug that inhibits the P2Y12which is a subtype of adenosine diphosphate (ADP)receptor.

It is a potent , direct-acting oral agent and it is reversibly binding P2Y12 receptors antagonist unlike the irreversible agents as clopidogrel, prasugrel, ticlopidine.

In 2011, the U.S. Food and Drug Administration (FDA) approved the blood-thinning drug (ticagrelor) to treat acute coronary syndromes, and in 2015, it approved it as long-term treatment in patient with history of heart attack.

In 2018, the American Heart Association ( AHA ) and American stroke Association (ASA) Guidelines for the Early Management of Patients with Acute Ischemic Stroke stated that, ticagrelor was not found to be superior to aspirin. However, because there were no significant safety differences, ticagrelor may be a reasonable alternative in stroke patients who have a contraindication to aspirin.

Aspirin overall reduces the risk of major vascular events by 13% Moreover, the risk of hemorrhagic events limits the use of aspirin in this setting, so the investigators aim at examining the hemorrhagic risks associated with use of loading Ticagrelor 180 ml within 9 hours of 1st ever acute ischemic stroke and compare the neurological outcomes in two groups of patients with 1st ever acute ischemic stroke receiving within 9 hours either Aspirin(300 mg (4 tablets of 75 mg) as a single loading oral dose, and will then be commenced on 300 mg Aspirin daily for 2 weeks then 75 mg daily after that for 3 months and the other received 180 mg ticagrelor (2 tablets of 90 mg) as a single loading oral dose, and continue on 180 mg ticagrelor (1 tablet of 90 mg every 12 hours) for 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male & female patients will be included
2. Age between 18 - 75 years
3. First ever presentation with acute ischemic stroke.Previous transient ischemic attacks (TIA's) are not excluding
4. Ictus to drug time does not to exceed 9 hours.

Exclusion Criteria

1. Patient eligible for recombinant tissue plasminogen activator (rTPA)
2. patients with( national institute of health stroke scale (NIHSS) below 3 or above 25
3. patients with active malignancy
4. patients with major surgery in past 3 months
5. patients with known allergy to study drugs
6. patients with acute myocardial infarction in past 6 months
7. patients known to suffer from multiple sclerosis or epilepsy
8. pregnancy or lactation
9. patients with history of head trauma with residual neurological deficits
10. patients on regular ticagrelol in past week
11. patients with international normalized ratio (INR) more than 1.3 or prothrombin time (PT) more than 18
12. patients with venous thrombosis
13. patients with platelet count less than 100000 or white blood cells (WBCs) less than 3000 or hematocrit value less than 0.25
14. blood glucose less than 50 mg/DL or more than 400

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
hemorrhagic transformation of infarction within 48 hours of loading anti platelet in each group | 48 hours
  hemorrhagic transformation detected by brain imaging CT and/or MRI brain will be done after 2 days of onset
amount of peripheral bleeding within 48 hours of loading anti platelet in each group | 48 hours
  amount of peripheral bleeding measured in milliliter in each group
frequency of peripheral bleeding within 48 hours of loading anti platelet in each group | 48 hours
  amount of peripheral bleeding measured as ( time per day )

SECONDARY OUTCOMES:
difference between National institute of health stroke scale scores on admission and after one week in each group | one week or discharge
  National institute of health stroke scale ( NIHSS) difference between score on admission and after one week: we consider favorable outcome if there is decrease in NIHSS by 4 points or more this scale ranges from 0 to 42 . the higher the value the worse outcome with the following values: 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
Modified Rankin scale in each group | after one week and after 3 months
  Modified Rankin Scale (MRS): assessed at the end of 3 months , the higher the value the worse the outcome , MRS has following values :
  0 = No symptoms at all
  * 1= No significant disability despite symptoms
  * 2= Slight disability
  * 3= Moderate disability
  * 4= Moderately severe disability
  * 5= Severe disability; bedridden
  * 6= Dead we consider favorable mRS if it was 2 or less
Mortality in each group | 3 months
  Timing and cause of death will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Hani Mohamed M Aref, MD, Study Chair — neuropsychiatry department Ain shams faculty of medicine; Hala M Elkhawas, MD, Study Director — neuropsychiatry department Ain shams faculty of medicine; Ahmed I Elbassiouny, MD, Study Director — neuropsychiatry department Ain shams faculty of medicine; Tamer M Roushdy, MD, Study Director — neuropsychiatry department Ain shams faculty of medicine; Hossam S Mohammed, MD, Study Director — neuropsychiatry department Ain shams faculty of medicine; Mohamed Zeinhom M Gomaa, M.Sc., Principal Investigator — neuropsychiatry department Kafrelsheikh faculty of medicine
Locations (1):
- Neuropsychiatry department Kafrelsheikh university hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the individual participant data for all primary and secondary outcomes measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available after 6 months of study completion
Access Criteria: data access requests will be reviewed by an external independent review panel , requestors will be required to sign a data access agreement

REFERENCES:
- [Result] Johnston SC, Amarenco P, Albers GW, Denison H, Easton JD, Evans SR, Held P, Jonasson J, Minematsu K, Molina CA, Wang Y, Wong KS; SOCRATES Steering Committee and Investigators. Ticagrelor versus Aspirin in Acute Stroke or Transient Ischemic Attack. N Engl J Med. 2016 Jul 7;375(1):35-43. doi: 10.1056/NEJMoa1603060. Epub 2016 May 10. PMID 27160892
- [Derived] Aref HM, El-Khawas H, Elbassiouny A, Shokri HM, Zeinhom MG, Roushdy TM. A randomized pilot study of the efficacy and safety of loading ticagrelor in acute ischemic stroke. Neurol Sci. 2023 Feb;44(2):765-771. doi: 10.1007/s10072-022-06525-7. Epub 2022 Nov 30. PMID 36446950
- [Derived] Zeinhom MG, Aref HM, El-Khawas H, Roushdy TM, Shokri HM, Elbassiouny A. A pilot study of the ticagrelor role in ischemic stroke secondary prevention. Eur Neurol. 2022;85(1):50-55. doi: 10.1159/000518786. Epub 2021 Aug 30. PMID 34515113
- See also: https://www.ncbi.nlm.nih.gov/pubmed/27160892 — https://www.ncbi.nlm.nih.gov/pubmed/27160892